CLINICAL TRIAL: NCT06795178
Title: A Global, Phase 3, Open-Label, Single Arm Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of FP-014, 11.25 mg (Triptorelin Mesylate Injection, 11.25 mg) in Patients With Advanced Prostate Cancer (KATANA E3M)
Brief Title: Efficacy, Safety, and Pharmacokinetics of FP-014, 11.25 mg in Patients With Advanced Prostate Cancer
Acronym: KATANA E3M
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons not safety related.
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP014C-24-001
Record Dates: First submitted 2025-01-22; First posted 2025-01-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FP-014, 11.25 mg (Experimental): Each patient will receive 2 single doses of FP-014, 11.25 mg administered as SC injections. The two injections of the study drug will be administered 12 weeks apart; one injection at Baseline (Visit 2/Day 0/Week 1), and one at Visit 13 (Day 84/Week 12) to achieve castrate serum testosterone level (< 50 ng/dL).
  Interventions: Drug: FP-014

INTERVENTIONS:
Drug: FP-014 — 11.25 mg in a prefilled, ready-to-use, long-acting formulation
  Other Names: Triptorelin Mesylate

SUMMARY:
This is a study in male patients with advanced prostate cancer who are eligible for androgen ablation therapy. The study duration will be up to 26 weeks.

Eligibility will be assessed during a screening period of up to 28 days. Up to 2 doses of a long-acting FP-014, 11.25 mg formulation will be given to the patients by separate SC injections 12 weeks apart in an unblinded manner. The first dose of FP-014, 11.25 mg, will be administered on Day 0 (Visit 2/Week 1). When patients have tolerated the first dose of FP-014, 11.25 mg and have achieved castrate levels of serum testosterone, a second dose will be administered on Day 84 (Visit 13/Week 12) to achieve castrate levels of serum testosterone concentrations (< 50 ng/dL). Patients will be followed for efficacy, safety, tolerability, and ancillary clinical and laboratory markers for an additional 12-week observation period (Day 168/Week 24/ Visit 22).

Blood samples will be collected at Baseline (Day 0/Week 1) at least 30 minutes before the first FP-014, 11.25 mg administration, immediately thereafter and at specified time points through Day 168 (Week 24) to determine pharmacokinetic (PK) (triptorelin) and pharmacodynamic (PD) (testosterone, PSA, and LH) profiles.

DETAILED DESCRIPTION:
This is a study in male patients with advanced prostate cancer who are eligible for androgen ablation therapy. The study duration will be up to 26 weeks.

Eligibility will be assessed during a screening period of up to 28 days. Up to 2 doses of a long-acting FP-014, 11.25 mg formulation will be given to the patients by separate SC injections 12 weeks apart in an unblinded manner. The first dose of FP-014, 11.25 mg, will be administered on Day 0 (Visit 2/Week 1). When patients have tolerated the first dose of FP-014, 11.25 mg and have achieved castrate levels of serum testosterone, a second dose will be administered on Day 84 (Visit 13/Week 12) to achieve castrate levels of serum testosterone concentrations (< 50 ng/dL). Patients will be followed for efficacy, safety, tolerability, and ancillary clinical and laboratory markers for an additional 12-week observation period (Day 168/Week 24/ Visit 22).

Blood samples will be collected at Baseline (Day 0/Week 1) at least 30 minutes before the first FP-014, 11.25 mg administration, immediately thereafter and at specified time points through Day 168 (Week 24) to determine pharmacokinetic (PK) (triptorelin) and pharmacodynamic (PD) (testosterone, PSA, and LH) profiles.

To evaluate the sustained castration testosterone level after two administrations of FP-014, 11.25 mg, the first 30 enrolled patients will be considered as a subset for safety and PK assessments. Furthermore, these 30 patients will be extended for another 2 weeks post Day 168 (Day 182 ± 2 days/Week 26/Visit 23) to obtain the extended PK/PD profiles of serum triptorelin mesylate and testosterone levels.

To evaluate the sustained castration testosterone level after two administrations of FP-014, 11.25 mg, the first 30 enrolled patients will be considered as a subset for safety and PK assessments. Furthermore, these 30 patients will be extended for another 2 weeks post Day 168 (Day 182 ± 2 days/Week 26/Visit 23) to obtain the extended PK/PD profiles of serum triptorelin mesylate and testosterone levels.

The efficacy assessments will be performed in both Intent-to-Treat (ITT) and Per-Protocol (PP) populations. Efficacy assessment will include the percentage of patients who reached the castrate levels (< 50 ng/dL) of serum testosterone on Day 28 (± 2 days; Week 4) post the first dosing of FP-014, 11.25 mg. Furthermore, the effect of FP-014, 11.25 mg on serum levels of PSA, and LH will be assessed post the first and the second dosing of FP-014, 11.25 mg, respectively. Urinary tract signs and symptoms will be evaluated for efficacy using the International Prostate Symptom Score (I-PSS) and will be recorded in the electronic case report forms (eCRFs). The acute-on-chronic (surge) effect of serum testosterone and LH levels will also be monitored in all patients. In addition, the impact of FP-014, 11.25 mg, on the percentage (rate) of patients with PSA relapse, on the percentage of patients that achieves normal serum PSA level, and on the percentage of patients with an enhanced serum testosterone concentration suppression (< 20 ng/dL) will be determined at the end of study.

All treatment emergent adverse events (TEAEs), including AEs of interest (AEoI), that occur during the study period and serious adverse events (SAEs) that occur during the study period will be recorded in the electronic case report forms (eCRFs) and followed until they are resolved or considered stable. In addition, all SAEs will be recorded and reported as required by local and international regulatory requirements.

Other safety assessments and their results, including safety clinical laboratory parameters, vital signs, physical examination, resting 12-lead electrocardiogram (ECG), injection site reactions and bone pain assessed using visual analog scale (VAS) will also be recorded in the eCRF.

Patients who discontinue early should be encouraged to remain in the study for safety evaluations.

A Data Safety Monitoring Board (DSMB) composed of independent experts will review available safety results every 3 months, and on an ad hoc basis if deemed necessary, from the moment onwards when one month data is available from approximately 5% of enrolled patients until the last patient completes the study. The composition and responsibilities of the DSMB will be defined in a separate DSMB charter.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 18 years old at Screening.
2. Histologically confirmed carcinoma of the prostate at the time of Screening.
3. Metastatic or biochemically recurrent prostate cancer disease at Screening.
4. Patient agrees to use male contraceptive methods during the study.
5. In the Investigator's opinion, the patient understands the nature of the study and any hazards of participation, communicates satisfactorily with the Investigator, and is able to participate in and comply with the requirements of the entire protocol.
6. Patients judged by the attending physician and/or Principal Investigator to be a candidate for androgen ablation therapy.
7. Patients who are able to tolerate androgen ablation therapy but are considered unable to tolerate androgen receptor pathway inhibitors.
8. ECOG Performance Status score ≤ 2 and life expectancy of at least 18 months at Screening.
9. Baseline morning serum testosterone level > 150 ng/dL at Screening.
10. Laboratory values at Screening:

    * Absolute neutrophil count ≥ 1,500 cells/μL;
    * Platelets ≥ 100,000 cells/μL;
    * Hemoglobin ≥ 10 gm/dL;
    * Total bilirubin ≤ 1.5 × upper limit of normal (ULN);
    * AST ≤ 2.5 × ULN;
    * ALT ≤ 2.5 × ULN;
    * Creatinine Clearance ≥ 30 mL/min or estimated Glomerular Filtration Rate (eGFR) > 30 mL/min/1.73 m2 or evidence of acute kidney injury;
    * Lipid profile within the acceptable range according to the Investigator's opinion;
    * Serum glucose within the acceptable range according to the Investigator's opinion;
    * HbA1c within the acceptable range according to the Investigator's opinion;
    * Clinical chemistries (K, Na, Mg, Ca, and P) within the acceptable range according to the Investigator's opinion;
    * Normal urinalysis results:

      * ed blood cells (RBCs) ≤ 3 RBCs/hpf;
      * white blood cells (WBCs) ≤ 5 WBCs/hpf;
      * nitrate: negative;
      * glucose: <0.1 g/dL in patients without diabetes mellitus Type II and < 1.0 g/dL in patients with diabetes mellitus Type II.

Exclusion Criteria:

1. Receipt of chemotherapy, immunotherapy, cryotherapy, radiotherapy, or anti-androgen therapy within 8 weeks prior to Screening, for treatment of carcinoma of the prostate.
2. Receipt of any luteinizing hormone-releasing hormone (LH-RH) suppressive therapy within 6 months of the screening visit.
3. Receipt of any vaccination (including influenza) within 2 weeks of the screening visit.
4. History of blood donation within 2 months of the screening visit.
5. History of anaphylaxis to any LH-RH analogues.
6. Contraindication to triptorelin or an LH-RH agonist as indicated on the package labeling.
7. Previous exposure to triptorelin mesylate.
8. Major surgery, including any prostatic surgery (excluding prostatic biopsy), within 4 weeks of the screening visit.
9. History of bilateral orchiectomy, adrenalectomy, or hypophysectomy.
10. History of clinical and radiographic evidence of central nervous system dysfunction.
11. Spinal cord metastases and patients at risk for spinal cord compression.
12. Clinical evidence of uncontrolled active urinary tract obstruction and patients at risk for urinary obstruction.
13. Clinically significant abnormal ECG at Screening and/or history of clinically significant ECG.
14. Cardiovascular disease that is clinically significant as judged by the Investigator.
15. History of uncontrolled diabetes, HbA1C >9.5%, urine glycosuria >1.0 g/dl, or presence of diabetic ketoacidosis.
16. History of liver dysfunction, including patients with moderate (Child-Pugh B) or severe (Child-Pugh C) impairment or disordered coagulation.
17. End-stage renal diseases on peritoneal dialysis or hemodialysis.
18. History or presence of hypogonadism; or receipt of exogenous testosterone supplementation within 6 months of screening visit.
19. Use of systemic corticosteroids at a dose > 10 mg/day at Screening.
20. Use of 5-alpha reductase inhibitor within the last 6 months of screening visit.
21. Use of any over-the-counter (OTC) medication within 4 weeks of the screening visit, except for those listed as permitted concomitant treatment.
22. History of drug and/or alcohol abuse within 6 months of screening visit.
23. Use of any investigational agent within 4 weeks of the screening visit.
24. Use of any therapeutics with strong inhibitors and strong inducers of CYP3A4 or CYP2C8 [e.g., rifampicin, ketoconazole, phenytoin, ritonavir, macrolide antibiotics (e.g. telithromycin)] at the time of Screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints | Week 4 (Day 28 ± 1 day) through Week 24 (Day 168 ± 5 days).
  The percentage of patients with a serum testosterone concentration suppressed to castrate levels (< 50 ng/dL) by Week 4 (Day 28 ± 1 day) following the first SC injection of FP-014 (11.25 mg).
  The percentage of patients with serum testosterone concentration suppressed to castrate levels (< 50 ng/dL)

SECONDARY OUTCOMES:
Secondary Endpoints | Week 24/End of Study (EOS) (Day 168 ± 5 days).
  The mean acute-on-chronic (surge) changes in serum testosterone and LH levels prior to the second injection through 48-72 hours after the second injection of FP-014, 11.25 mg.
  The mean change of serum LH levels
Secondary Endpoints | Baseline to Week 24/EOS (Day 168 ± 5 days).
  The mean change of serum PSA levels
Secondary Endpoints | Week 24/EOS (Day 168 ± 5 days)/Week 24/EOS (Day 168 ± 5 days).
  The percentage of patients with:
  . PSA relapse (defined as an increase in serum PSA of > 50% PSA nadir by Week 24/EOS (Day 168 ± 5 days) after achieving serum PSA level ≤ 4 ng/mL post administration of FP-014, 11.25 mg.
  Within normal limit serum PSA level (≤ 4 ng/mL) by Week 24/EOS (Day 168 ± 5 days).
Secondary Endpoints | Week 4 (Day 28 ± 1 day) and at Week 24/EOS (Day 168 ± 5 days)
  The percentage of patients with enhanced serum testosterone concentration suppression to < 20 ng/dL
Secondary Endpoints | Baseline to Week 24/EOS (Day 168 ± 5 days).
  Urinary signs and symptoms, i.e. a patient-reported outcome (PRO) assessed by the total score of the International Prostate Symptom Score (I-PSS) sheet (Range 0-35 with 35 being the worst symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Whitaker, BSN, MS, MBA, Study Director — Foresee Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No